CLINICAL TRIAL: NCT04769375
Title: Investigation of the Effect of Gestational Diabetes Mellitus on the Pelvic Girdle Pain and Symptom Severity in Pregnant Women
Brief Title: Pelvic Girdle Pain in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 31
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-02

CONDITIONS: Gestational Diabetes; Pelvic Girdle Pain; Pregnant Woman
Keywords: gestational diabetes mellitus, pregnancy pelvic girdle pain
MeSH Terms: conditions — Diabetes, Gestational; Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Pregnant women diagnosed with GDM (first pregnancy): This group will consist of women with gestational diabetes mellitus according to routine control tests in their first pregnancy.
  Interventions: Other: Evaluation of pain; Other: Application of pelvic girdle pain tests; Other: Application of pelvic girdle questionnaire
- Group 2:Pregnant women diagnosed with GDM (2nd or 3rd pregnancy): This group will consist of women with gestational diabetes mellitus according to routine control tests in their second or third pregnancy.
  Interventions: Other: Evaluation of pain; Other: Application of pelvic girdle pain tests; Other: Application of pelvic girdle questionnaire
- Group 3: Healthy pregnant women (first pregnancy): This group will consist of women who do not have gestational diabetes mellitus according to routine control tests in their first pregnancy.
  Interventions: Other: Evaluation of pain; Other: Application of pelvic girdle pain tests; Other: Application of pelvic girdle questionnaire
- Group 4:Healthy pregnant women (2nd or 3rd pregnancy): This group will consist of women who do not have gestational diabetes mellitus according to routine control tests in their second or third pregnancy.
  Interventions: Other: Evaluation of pain; Other: Application of pelvic girdle pain tests; Other: Application of pelvic girdle questionnaire

INTERVENTIONS:
Other: Evaluation of pain — The presence of pain localization pelvic girdle pain will be questioned in the body chart. Inaddition to this, the level of the pelvic girdle pain will be evaluated by visual analog scale.
Other: Application of pelvic girdle pain tests — The tests will be applied sequentially to investigate the presence and severity of the pain (Tests: Posterior Pelvic Pain Provocation, Patriarch FABER, Long Dorsal Sacroiliac Ligament Pain Provocation, Simpsis Palpation, Modified Trendelenburg and Active Straight Leg Raise)
Other: Application of pelvic girdle questionnaire — Pelvic girdle questionnaire will be filled by pregnant women with pelvic girdle pain.

SUMMARY:
Pelvic girdle pain and gestational diabetes mellitus are experienced in similar trimesters of pregnancy. The aim of this study is to examine the effect of gestational diabetes mellitus on the occurrence of pelvic girdle pain and the severity of symptoms of pelvic girdle pain in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women diagnosed with GDM in the 2nd and 3rd trimesters Pregnant women without GDM diagnosis in 2nd and 3rd trimester First pregnancy Second or third pregnancy 20-40 years old

Exclusion Criteria:

Diabetes mellitus before pregnancy The presence of an orthopedic or neurological problem that may cause musculoskeletal disorder and biomechanical sequence deviations from normal Pre-pregnancy chronic lumbar-pelvic pain description History of spine, pelvis or lower extremity surgery or fracture in the past 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: Pegnant women with gestational diabetes mellitus (first pregnancy) Pegnant women with gestational diabetes mellitus (second or third pregnancy) Pegnant women without gestational diabetes mellitus (first pregnancy) Pegnant women without gestational diabetes mellitus (second or third pregnancy)
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | Baseline
  Measuring of the presence of pain and severity level of pain with body chart and vısual analog scale
Evaluation of test of pelvic girdle | Baseline
  Measuring of the presence of pain and severity level of pain with pelvic girdle provocation and palpation tests
Evaluation of pelvic girdle questionnaire | Baseline
  Measuring of the pelvic girdle questionnaire (PGQ) in pregnant women with pelvic girdle pain

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Result] Eberhard-Gran M, Eskild A. Diabetes mellitus and pelvic girdle syndrome in pregnancy--is there an association? Acta Obstet Gynecol Scand. 2008;87(10):1015-9. doi: 10.1080/00016340802345944. PMID 18763174
- [Result] Eivazi M, Abadi L. Low back pain in diabetes mellitus and importance of preventive approach. Health Promot Perspect. 2012 Jul 1;2(1):80-8. doi: 10.5681/hpp.2012.010. eCollection 2012. PMID 24688921
- [Result] Plows JF, Stanley JL, Baker PN, Reynolds CM, Vickers MH. The Pathophysiology of Gestational Diabetes Mellitus. Int J Mol Sci. 2018 Oct 26;19(11):3342. doi: 10.3390/ijms19113342. PMID 30373146
- [Result] Wuytack F, O'Donovan M. Outcomes and outcomes measurements used in intervention studies of pelvic girdle pain and lumbopelvic pain: a systematic review. Chiropr Man Therap. 2019 Nov 5;27:62. doi: 10.1186/s12998-019-0279-2. eCollection 2019. PMID 31700607
- [Result] Stuge B, Garratt A, Krogstad Jenssen H, Grotle M. The pelvic girdle questionnaire: a condition-specific instrument for assessing activity limitations and symptoms in people with pelvic girdle pain. Phys Ther. 2011 Jul;91(7):1096-108. doi: 10.2522/ptj.20100357. Epub 2011 May 19. PMID 21596959
- [Result] Palsson TS, Beales D, Slater H, O'Sullivan P, Graven-Nielsen T. Pregnancy is characterized by widespread deep-tissue hypersensitivity independent of lumbopelvic pain intensity, a facilitated response to manual orthopedic tests, and poorer self-reported health. J Pain. 2015 Mar;16(3):270-82. doi: 10.1016/j.jpain.2014.12.002. Epub 2014 Dec 23. PMID 25540938
- [Result] Molsted S, Tribler J, Snorgaard O. Musculoskeletal pain in patients with type 2 diabetes. Diabetes Res Clin Pract. 2012 May;96(2):135-40. doi: 10.1016/j.diabres.2011.12.022. Epub 2012 Jan 12. PMID 22244365
- [Result] Martins RF, Pinto e Silva JL. Treatment of pregnancy-related lumbar and pelvic girdle pain by the yoga method: a randomized controlled study. J Altern Complement Med. 2014 Jan;20(1):24-31. doi: 10.1089/acm.2012.0715. Epub 2013 Mar 18. PMID 23506189